CLINICAL TRIAL: NCT06236165
Title: Clinical Study Evaluating Efficacy, Safety and Molecular Mechanism of N-acetylcysteine Supplementation in Patients With Hepatic and Post Hepatic Jaundice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samah Hussein Mohamed, Master degree in Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00543/2024
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-01

CONDITIONS: Hepatic and Post Hepatic Jaundice
Keywords: Jaundice; N-acetylcysteine; TAC; TNF-α; Bilirubin
MeSH Terms: conditions — Jaundice | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): 22 patients who will receive supportive treatment for jaundice only, for 3 months.
- NAC arm (Experimental): 22 patients who will receive oral N-acetylcysteine 600 mg twice daily in addition to supportive treatment, for 3 months.
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Patients will receive oral N-acetylcysteine 600 mg twice daily in addition to supportive treatment, for 3 months.
  Arms: NAC arm

SUMMARY:
Investigating the efficacy, safety, and molecular mechanism of N-acetylcysteine supplementation in improving elevated direct bilirubin level and liver function tests in patients with hepatic and post-hepatic jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-70 years old.
* Patients diagnosed with jaundice and increased level direct bilirubin ≥ 3 mg/dL.

Exclusion Criteria:

* Pregnancy.
* Nursing mothers.
* Patients with increased indirect bilirubin level.
* Patients who have Gilbert syndrome or Crigler Najjar syndrome.
* Patients with Child Paugh C score (10-15 point).
* History of known hypersensitivity to N-acetylcysteine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Change in total antioxidant capacity (TAC) level | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Assessment of total antioxidant capacity (TAC) level by ELISA Kits according to manufacturer's instructions.
Change in tumor necrosis factor alpha (TNF-α) | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Assessment of tumor necrosis factor alpha (TNF-α) level by ELISA Kits according to manufacturer's instructions

SECONDARY OUTCOMES:
Adverse events and toxicity | 3 months.
  Adverse events and toxicity will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
Follow up of liver function | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  measurement of alanine transaminase (ALT) and aspartate transaminase (AST) both in U/L from blood samples will be assessed for all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Samah Hussein, Principal Investigator — Tanta University
Locations (1):
- Faculty of Pharmacy, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No